CLINICAL TRIAL: NCT02104609
Title: Pharmacokinetics of the Levonorgestrel-only Emergency Contraception Regimen in Normal-weight, Obese and Extremely Obese Users: a Pilot Study
Brief Title: Effects of Obesity on Pharmacokinetics of the Levonorgestrel Emergency Contraceptive Pill
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Melissa Natavio, Asst. Professor, University of Southern California
Other Study IDs: HS-12-00602
Record Dates: First submitted 2014-03-25; First posted 2014-04-04 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Obesity
Keywords: Obesity; Emergency contraception; Levonorgestrel emergency contraception
MeSH Terms: conditions — Obesity | interventions — Levonorgestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Normal weight women: Levonorgestrel 1.5mg by mouth once
  Interventions: Drug: Levonorgestrel 1.5mg by mouth once
- Obese women: Levonorgestrel 1.5mg by mouth once
  Interventions: Drug: Levonorgestrel 1.5mg by mouth once
- Extremely obese women: Levonorgestrel 1.5mg by mouth once
  Interventions: Drug: Levonorgestrel 1.5mg by mouth once

INTERVENTIONS:
Drug: Levonorgestrel 1.5mg by mouth once — Levonorgestrel 1.5mg by mouth given on menstrual cycle day 8
  Other Names: Plan B One Step; Next Choice One Dose

SUMMARY:
The purpose of this study is to determine the effects of obesity on the pharmacokinetics of the levonorgestrel (LNG) only emergency contraceptive (EC) regimen and on markers of ovulation

Primary hypothesis:

1) Obese users of LNG-EC have a pharmacokinetic profile that is consistent with a larger volume of distribution of LNG.

Secondary hypothesis:

1. Alterations in these pharmacokinetic parameters of the LNG-EC regimen in obese women affect the primary mechanism of action, which is inhibition of ovulation.
2. Obesity may affect other factors that alter levels of LNG, such as sex-hormone binding globulin (SHBG) and albumin, which bind LNG and potentially lowers the amount of free LNG.

ELIGIBILITY:
Inclusion Criteria:

* Women between ages 18-35 years

  * Regular menstrual cycles (24-35 days) for the past 2 months
  * Ovulatory at defined by midluteal progesterone level >3 ng/mL (Day 18-25)
  * Belongs to one of the following categories: normal weight (BMI = 18.5-24.9 kg/m2), obese (BMI = 30-39.9 kg/m2) or extremely obese (BMI ≥ 40 kg/m2)
  * Participant has no intention of or desire to conceive (e.g., active attempt to become pregnant or in vitro fertilization) for the duration of the study
  * Participant agrees to consistently use an effective method of nonhormonal contraception throughout the duration of study, which could include: condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, non-hormonal intra-uterine devise (IUD), or sterilization.
  * Able to give informed consent

Exclusion Criteria:

* • Known renal or liver disease

  * Known pituitary disorder
  * Known adrenal disorder
  * Known thyroid disorder
  * Use of medication known to alter the cytochrome P450 system
  * Use of depot-medroxyprogesterone acetate in the previous 6 months or any other hormonal contraceptive in the previous 3 months
  * Currently breastfeeding
  * Pregnant
  * Pregnancy in the prior month
  * Known allergy to medication
  * Other specific contraindications to LNG EC

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Non-smoking women between ages 18-35 years with regular menstrual cycles (24-35 days) will be enrolled, to include 10 normal weight (BMI = 18.5-24.9 kg/m2) women, 10 obese (BMI = 30-39.9 kg/m2) and 10 extremely obese (BMI ≥ 40 kg/m2) women
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2013-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) | Time 0, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 hours

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) | 0, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 hours
Minimum concentration (Cmin) | Time 0, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 hours
Area under the concentration time-curve (AUC) | Time 0, 1, 2, 3, 4, 6, 8, 12, 6, 24, 48, 72 hrs

CONTACTS AND LOCATIONS:
Overall Officials: M Natavio, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States